CLINICAL TRIAL: NCT05211323
Title: A Randomized Phase II Trial Evaluating Chemotherapy Plus Atezolizumab vs Chemotherapy Plus Bevacizumab and Atezolizumab in Advanced Combined Hepatocellular Carcinoma-Cholangiocarcinoma
Brief Title: A Study to Determine Whether Chemotherapy and Atezolizumab is Better Than Chemotherapy, Bevacizumab and Atezolizumab in Patients With Advanced Liver Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2022-00151; NCI-2022-00151 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); EA2205 (Other: ECOG-ACRIN Cancer Research Group); EA2205 (Other: CTEP); U10CA180820 (NIH)
Record Dates: First submitted 2022-01-22; First posted 2022-01-27 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Combined Hepatocellular Carcinoma and Cholangiocarcinoma; Stage III Liver Cancer; Stage IV Liver Cancer
MeSH Terms: conditions — Liver Neoplasms | interventions — atezolizumab; Bevacizumab; Immunoglobulin G; Disulfides; Specimen Handling; Cisplatin; 1,2-diaminocyclohexaneplatinum II citrate; Platinum; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (atezolizumab, bevacizumab, gemcitabine, cisplatin) (Experimental): Patients receive atezolizumab IV over 30-60 minutes on day 1, bevacizumab IV over 30-90 minutes on day 1, gemcitabine IV over 30 minutes on days 1 and 8, and cisplatin IV on days 1 and 8. Cycles repeats every 21 days in the absence of disease progression or unacceptable toxicity. Patients undergo CT or MRI throughout the trial. Patients undergo blood specimen collection on study.
  Interventions: Biological: Atezolizumab; Biological: Bevacizumab; Procedure: Biospecimen Collection; Drug: Cisplatin; Procedure: Computed Tomography; Procedure: Conventional Magnetic Resonance Imaging; Drug: Gemcitabine Hydrochloride
- Arm B (atezolizumab, gemcitabine, cisplatin) (Active Comparator): Patients receive atezolizumab IV over 30-60 minutes on day 1, and gemcitabine IV over 30 minutes and cisplatin IV on days 1 and 8. Cycles repeats every 21 days in the absence of disease progression or unacceptable toxicity. Patients undergo CT or magnetic resonance imaging MRI throughout the trial. Patients undergo blood specimen collection on study.
  Interventions: Biological: Atezolizumab; Procedure: Biospecimen Collection; Drug: Cisplatin; Procedure: Computed Tomography; Procedure: Conventional Magnetic Resonance Imaging; Drug: Gemcitabine Hydrochloride

INTERVENTIONS:
Biological: Atezolizumab — Given IV
  Other Names: MPDL 3280A; MPDL 328OA; MPDL-3280A; MPDL3280A; MPDL328OA; RG 7446; RG-7446; RG7446; RO 5541267; RO-5541267; RO5541267; Tecentriq
Biological: Bevacizumab — Given IV
  Other Names: ABP 215; ABP-215; ABP215; Alymsys; Anti-VEGF; Anti-VEGF Humanized Monoclonal Antibody; Anti-VEGF Monoclonal Antibody SIBP04; Anti-VEGF rhuMAb; Avastin; Avzivi; Aybintio; BAT 1706; BAT-1706; BAT1706; BAT1706 Biosimilar; Bevacizumab awwb; Bevacizumab Biosimilar ABP 215; Bevacizumab Biosimilar BAT1706; Bevacizumab Biosimilar BEVZ92; Bevacizumab Biosimilar BI 695502; Bevacizumab Biosimilar CBT 124; Bevacizumab Biosimilar CT-P16; Bevacizumab Biosimilar FKB238; Bevacizumab Biosimilar GB-222; Bevacizumab Biosimilar HD204; Bevacizumab Biosimilar HLX04; Bevacizumab Biosimilar IBI305; Bevacizumab Biosimilar LY01008; Bevacizumab Biosimilar MB02; Bevacizumab Biosimilar MIL60; Bevacizumab Biosimilar Mvasi; Bevacizumab Biosimilar MYL-1402O; Bevacizumab Biosimilar QL 1101; Bevacizumab Biosimilar QL1101; Bevacizumab Biosimilar RPH-001; Bevacizumab Biosimilar SCT501; Bevacizumab Biosimilar Zirabev; Bevacizumab-adcd; Bevacizumab-awwb; Bevacizumab-aybi; Bevacizumab-bvzr; Bevacizumab-equi; Bevacizumab-maly; Bevacizumab-onbe; Bevacizumab-tnjn; BP102; BP102 Biosimilar; CT P16; CT-P16; CTP16; Equidacent; FKB 238; FKB-238; FKB238; HD204; Immunoglobulin G1 (Human-Mouse Monoclonal rhuMab-VEGF Gamma-Chain Anti-Human Vascular Endothelial Growth Factor), Disulfide With Human-Mouse Monoclonal rhuMab-VEGF Light Chain, Dimer; MB 02; MB-02; MB02; Mvasi; MYL-1402O; Onbevzi; Oyavas; PF 06439535; PF-06439535; PF06439535; QL1101; Recombinant Humanized Anti-VEGF Monoclonal Antibody; rhuMab-VEGF; SCT501; SIBP 04; SIBP-04; SIBP04; Vegzelma; Zirabev
  Arms: Arm A (atezolizumab, bevacizumab, gemcitabine, cisplatin)
Procedure: Biospecimen Collection — Undergo blood specimen collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Drug: Cisplatin — Given IV
  Other Names: Abiplatin; Blastolem; Briplatin; CDDP; Cis-diammine-dichloroplatinum; Cis-diamminedichloridoplatinum; Cis-diamminedichloro Platinum (II); Cis-diamminedichloroplatinum; Cis-dichloroammine Platinum (II); Cis-platinous Diamine Dichloride; Cis-platinum; Cis-platinum II; Cis-platinum II Diamine Dichloride; Cismaplat; Cisplatina; Cisplatinum; Cisplatyl; Citoplatino; Citosin; Cysplatyna; DDP; Lederplatin; Metaplatin; Neoplatin; Peyrone's Chloride; Peyrone's Salt; Placis; Plastistil; Platamine; Platiblastin; Platiblastin-S; Platinex; Platinol; Platinol- AQ; Platinol-AQ; Platinol-AQ VHA Plus; Platinoxan; Platinum; Platinum Diamminodichloride; Platiran; Platistin; Platosin
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Procedure: Conventional Magnetic Resonance Imaging — Undergo MRI
  Other Names: Conventional MRI
Drug: Gemcitabine Hydrochloride — Given IV
  Other Names: dFdCyd; Difluorodeoxycytidine Hydrochloride; Gemcitabine HCI; Gemzar; LY 188011; LY-188011; LY188011

SUMMARY:
This phase II trial compares the effect of adding bevacizumab and atezolizumab to gemcitabine and cisplatin (chemotherapy) versus chemotherapy and atezolizumab in treating patients with liver cancer that cannot be removed by surgery (unresectable) or that may have spread from where it first started to nearby tissue, lymph nodes, or distant parts of the body (advanced). Immunotherapy with monoclonal antibodies, such as atezolizumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Bevacizumab is in a class of medications called antiangiogenic agents. It works by stopping the formation of blood vessels that bring oxygen and nutrients to tumor. This may slow the growth and spread of tumor. Chemotherapy drugs, such as gemcitabine and cisplatin, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving bevacizumab and atezolizumab with chemotherapy may kill more tumor cells in patients liver cancer than chemotherapy and atezolizumab.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate whether a quadruplet combined chemotherapy, immunotherapy, and anti-VEGF therapy improves progression-free survival (PFS), defined as time to progressive disease or death due to any cause as determined by the investigator using Response Evaluation Criteria in Solid Tumors (RECIST) version (v)1.1, compared to chemotherapy plus immunotherapy in patients with advanced combined hepatocellular carcinoma and cholangiocarcinoma (cHCC-CC).

SECONDARY OBJECTIVES:

I. To evaluate whether a quadruplet combined chemotherapy, immunotherapy, and anti-VEGF therapy improves objective response (OR), defined as a complete or partial response as determined by the investigator according to RECIST v1.1, compared to chemotherapy plus immunotherapy in patients with advanced cHCC-CC.

II. To evaluate whether a quadruplet combined chemotherapy, immunotherapy, and anti-VEGF therapy improves overall response (OS), and disease control rate as determined by the investigator using RECIST v1.1, compared to chemotherapy plus immunotherapy in patients with advanced cHCC-CC.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM A: Patients receive atezolizumab intravenously (IV) over 30-60 minutes on day 1, bevacizumab IV over 30-90 minutes on day 1, gemcitabine IV over 30 minutes on days 1 and 8, and cisplatin IV on days 1 and 8. Cycles repeats every 21 days in the absence of disease progression or unacceptable toxicity. Patients undergo computed tomography (CT) or magnetic resonance imaging (MRI) throughout the trial. Patients undergo blood specimen collection on study.

ARM B: Patients receive atezolizumab IV over 30-60 minutes on day 1, and gemcitabine IV over 30 minutes and cisplatin IV on days 1 and 8. Cycles repeats every 21 days in the absence of disease progression or unacceptable toxicity. Patients undergo CT or magnetic resonance imaging MRI throughout the trial. Patients undergo blood specimen collection on study.

After completion of study treatment, patients are followed up for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be >= 18 years of age
* Patient must have a histologically confirmed diagnosis of combined hepatocellular carcinoma-cholangiocarcinoma (cHCC-CC) at the local laboratory based on the 2019 World Health Organization (WHO) classification, including the classical type and intermediate cell carcinoma

  * The classical type defines primary liver carcinoma with unequivocal features of both HCC and CC differentiation within the same tumors on routine histopathology with hematoxylin and eosin stains regardless of the proportion of each histology observed
  * The intermediate cell carcinoma defines cancers with biphenotypic differentiation in which cells have a morphology intermediate between hepatocytes and cholangiocytes. Intermediate cell carcinoma may be associated with expression of both hepatocyte and cholangiocytic markers. Distinct HCC and CC arising in the same liver, fibrolamellar HCC, morphologically typical HCCs with only immunohistochemical expression of keratin or other cholangiocytic markers, or morphologically typical CCs with only immunohistochemical expression of hepatocytic markers will be excluded
  * NOTE: Local pathology review constitutes adequate documentation of histology for initial study enrollment and treatment
* Patient must have Eastern Cooperative Oncology Group (ECOG) performance status of 0-1
* Patient must have disease which is unresectable or metastatic
* Patient must not have any prior history of systemic therapy for advanced cHCC-CC. Prior adjuvant treatment composed of chemotherapy agents such as capecitabine or gemcitabine-based treatments are allowed if adjuvant treatment if at least 6 months have elapsed since completing chemotherapy at the time of enrollment
* Patient must be Child Pugh class A
* Patients with prior locoregional therapy are eligible provided the following are met:

  * Prior loco-regional therapy including surgical resection, chemoembolization, radiotherapy, or ablation was completed > 4 weeks prior to randomization
  * Treated target lesion has increased in size by > 25% or the target lesion was not treated with loco-regional therapy
  * Patients treated with palliative radiotherapy for symptoms must have completed radiotherapy > 7 days prior to randomization and the target lesion must not have been the treated lesion
* Patient must not be pregnant or breast-feeding due to the potential harm to an unborn fetus and possible risk for adverse events in nursing infants with the treatment regimens being used.

  * All patients of childbearing potential must have a blood test or urine study within 14 days prior to randomization to rule out pregnancy
  * A patient of childbearing potential is defined as anyone, regardless of sexual orientation or whether they have undergone tubal ligation, who meets the following criteria: 1) has achieved menarche at some point, 2) has not undergone a hysterectomy or bilateral oophorectomy; or 3) has not been naturally postmenopausal (amenorrhea following cancer therapy does not rule out childbearing potential) for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months)
* Patient must not expect to conceive or father children by abstaining from sexual intercourse or by using accepted and effective method(s) of contraception while on protocol treatment and for 6 months after the last dose of protocol treatment. Accepted and effective method(s) of contraception include those with a failure rate of < 1% per year including bilateral tubal ligation, male sterilization, hormonal contraceptives that inhibit ovluation, hormonal releasing intrauterine devices, and copper intrauterine devices. Periodic abstinence (e.g. calendar, ovulation, symptothermal, or postovulation methods) and withdrawal are not adequate methods of contraception
* Patient must have the ability to understand and the willingness to sign a written informed consent document. Patients with impaired decision-making capacity (IDMC) who have a legally authorized representative (LAR) or caregiver and/or family member available will also be considered eligible
* Leukocytes >= 3,000/mcL (must be obtained =< 14 days prior to protocol randomization)
* Absolute neutrophil count (ANC) >= 1,500/mcL (must be obtained =< 14 days prior to protocol randomization)
* Hemoglobin >= 9 g/dL (Patient may be transfused to meet this criterion) (must be obtained =< 14 days prior to protocol randomization)
* Platelets >= 80,000/mcL (must be obtained =< 14 days prior to protocol randomization)
* Total bilirubin =< 5 x institutional upper limit of normal (ULN) (must be obtained =< 14 days prior to protocol randomization)
* Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 5.0 x institutional ULN (must be obtained =< 14 days prior to protocol randomization)
* Creatinine =< 1.5 x institutional ULN (must be obtained =< 14 days prior to protocol randomization)
* International normalized ratio (INR) =< 1.5 x Institutional ULN (for patients not receiving anticoagulant therapy) (must be obtained =< 14 days prior to protocol randomization). For patients receiving therapeutic anticoagulation, the patient must be on a stable anticoagulant regimen
* Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months of randomization are eligible for this trial
* For patients with evidence of prior or active hepatitis B virus (HBV) infection (positive hepatitis B surface antigen [HBsAg] test and/or positive total hepatitis B virus core antibody [HBcAb] test at screening), the patient must be on suppressive therapy, for at least 2 weeks prior to randomization and willing to continue antiviral treatment for the length of the study
* Patient must not have new or progressive brain metastases (active brain metastases) or leptomeningeal disease
* Patients must not have laboratory evidence of active co-infection of HBV (positive HBsAg test) and hepatitis C virus (HCV) (detectable HCV ribonucleic acid [RNA]). Patients with a history of HCV infection but who are negative for HCV RNA by polymerase chain reaction (PCR) will be considered non-infected with HCV
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial
* Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, patients should be class 2B or better
* Patient must have measurable disease. Baseline measurements and evaluations of all sites of disease must be obtained within 4 weeks prior to randomization
* Patients with untreated or incompletely treated varices with bleeding or high-risk for bleeding must undergo an esophagogastroduodenoscopy (EGD), and all size of varices (small to large) must be assessed and treated per local standard of care prior to randomization. Patients who have undergone an EGD within 6 months of prior to randomization do not need to repeat the procedure
* Patient must not have had a prior allogenic bone marrow or solid organ transplant
* Patient must not have a history of idiopathic pulmonary fibrosis, organizing pneumonia, drug-induced pneumonitis, or idiopathic pneumonitis, or evidence of active pneumonitis on baseline chest computed tomography scan
* Patient must not have active or a history of autoimmune disease or immune deficiency, including, but not limited to, myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, antiphospholipid antibody syndrome, Wegener granulomatosis, Sjogren syndrome, Guillain-Barre syndrome, or multiple sclerosis, with the following exceptions:

  * Patients with a history of autoimmune-related hypothyroidism who are on thyroid-replacement hormone are eligible
  * Patients with controlled type 1 diabetes mellitus who are on an insulin regimen are eligible for the study
  * Patients with eczema, psoriasis, lichen simplex chronicus, or vitiligo with dermatologic manifestations only (e.g., patients with psoriatic arthritis are excluded) are eligible provided all of following conditions are met:

    * Rash must cover < 10% of body surface area
    * Disease is well controlled at baseline and requires only low-potency topical corticosteroids
    * There is no occurrence of acute exacerbations of the underlying condition requiring psoralen plus ultraviolet A radiation, methotrexate, retinoids, biologic agents, oral calcineurin inhibitors, or high-potency or oral corticosteroids
* Patient must not have received prior treatment with immune checkpoint blockade therapies, including anti-CTLA-4, anti-PD-1, and anti-PD-L1 therapeutic antibodies
* Patient must not be on treatment with systemic immunosuppressive medication (including, but not limited to, corticosteroids, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-TNF-alpha agents) within 2 weeks prior to randomization, or anticipate the need for systemic immunosuppressive medication during study treatment, with the following exceptions:

  * Patients who received acute, low-dose systemic immunosuppressant medication or a one-time pulse dose of systemic immunosuppressant medication (e.g., 48 hours of corticosteroids for a contrast allergy) are eligible
  * Patients who received mineralocorticoids (e.g., fludrocortisone), corticosteroids for chronic obstructive pulmonary disease (COPD) or asthma, or low-dose corticosteroids for orthostatic hypotension or adrenal insufficiency are eligible
* Patient must not have inadequately controlled arterial hypertension (defined as systolic blood pressure (BP) >= 150 mmHg and/or diastolic blood pressure > 100 mmHg) prior to randomization. Patients may be on antihypersensitive medications to meet and maintain this criteria
* Patient must not have significant vascular disease (e.g., aortic aneurysm requiring surgical repair or recent peripheral arterial thrombosis) within 6 months prior to randomization
* Patient may not have a history of abdominal or tracheoesophageal fistula, gastrointestinal (GI) perforation, or intra-abdominal abscess within 6 months prior to randomization
* Patient must not have any evidence of bleeding diathesis or significant coagulopathy (in the absence of therapeutic anticoagulation)
* Patient must not have uncontrolled tumor-related pain. Patients requiring pain medication must be on a stable regimen at the time of randomization

  * For patients with symptomatic lesions (e.g., bone metastases or metastases causing nerve impingement) amenable to palliative radiotherapy should be treated prior to randomization. Patients must be recovered from the effects of radiation prior to randomization. There is no required minimum recovery period
  * For patients with asymptomatic metastatic lesions that would likely cause functional deficits or intractable pain with further growth (e.g., epidural metastasis that is not currently associated with spinal cord compression) they must be considered for loco-regional therapy if appropriate prior to randomization
* Patient must not have uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures (once monthly or more frequently). Patients with indwelling catheters (e.g., PleurX) are allowed
* Patient must not have active tuberculosis
* Patient must not have undergone any major surgical procedure, other than for diagnosis, within 4 weeks prior to randomization, or have the anticipation of need for a major surgical procedure during the study
* Patient must not have any other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding that contraindicates the use of the agents used on this study, may affect the interpretation of the results, or may render the patient at high risk from treatment complications
* Patient must not have received any live, attenuated vaccines (e.g., FluMist [registered trademark]) within 4 weeks prior to randomization, during treatment with atezolizumab, and for 5 months after the last dose of atezolizumab
* Patient must not have received any treatment with investigational therapy within 28 days prior to randomization
* Patient must have not received treatment with systemic immunostimulatory agents (including, but not limited to, interferon and interleukin 2 [IL-2]) within 4 weeks or 5 half-lives of the drug (whichever is longer) prior to randomization
* Patients must not have a history of severe allergic anaphylactic reactions to chimeric or humanized antibodies or fusion proteins
* Patient must not have a known hypersensitivity to Chinese hamster ovary cell products or to any component of the atezolizumab formulation
* Patient must not have a known allergy or hypersensitivity to any component of the atezolizumab and bevacizumab formulation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2022-12-07 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) | From start of treatment until progression, assessed up to 3 years
  Defined as time to progressive disease or death due to any cause as determined by the investigator using Response Evaluation Criteria in Solid Tumors (RECIST) version (v)1.1. The null hypothesis of equality of PFS will be tested using a one-sided alternative favoring the quadruplet arm. The primary comparison will be via a one-sided log rank test.

SECONDARY OUTCOMES:
Objective response rate | Up to 3 years
  Defined as a complete or partial response as determined by the investigator according to RECIST v1.1. Will be tested using a Fisher's exact test at a one-sided significance level of 0.10.
Overall response rate | Up to 3 years
  Will be tested using a Fisher's exact test at a one-sided significance level of 0.10.

CONTACTS AND LOCATIONS:
Overall Officials: David Hsieh, Principal Investigator — ECOG-ACRIN Cancer Research Group
Locations (37):
- United States (37):
  - Sutter Auburn Faith Hospital, Auburn, California
  - Alta Bates Summit Medical Center-Herrick Campus, Berkeley, California
  - Palo Alto Medical Foundation-Fremont, Fremont, California
  - Memorial Medical Center, Modesto, California
  - Palo Alto Medical Foundation-Camino Division, Mountain View, California
  - Palo Alto Medical Foundation Health Care, Palo Alto, California
  - Sutter Roseville Medical Center, Roseville, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - California Pacific Medical Center-Pacific Campus, San Francisco, California
  - Palo Alto Medical Foundation-Santa Cruz, Santa Cruz, California
  - Palo Alto Medical Foundation-Sunnyvale, Sunnyvale, California
  - Sutter Solano Medical Center/Cancer Center, Vallejo, California
  - Carle at The Riverfront, Danville, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - The Carle Foundation Hospital, Urbana, Illinois
  - Memorial Hospital of South Bend, South Bend, Indiana
  - UI Health Care Mission Cancer and Blood - Ankeny Clinic, Ankeny, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - UI Health Care Mission Cancer and Blood - Des Moines Clinic, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - Miami Valley Hospital South, Centerville, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Premier Blood and Cancer Center, Dayton, Ohio
  - Miami Valley Hospital North, Dayton, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Miami Valley Cancer Care and Infusion, Greenville, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - Parkland Memorial Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Fort Worth, Fort Worth, Texas
  - UT Southwestern Clinical Center at Richardson/Plano, Richardson, Texas
  - VCU Massey Cancer Center at Stony Point, Richmond, Virginia
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - Marshfield Medical Center-EC Cancer Center, Eau Claire, Wisconsin
  - Marshfield Medical Center - Minocqua, Minocqua, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm

DOCUMENTS (1):
  • Informed Consent Form (2023-10-18): https://cdn.clinicaltrials.gov/large-docs/23/NCT05211323/ICF_000.pdf